CLINICAL TRIAL: NCT05813808
Title: Low-dose Computer Tomography in Follow-up of High Grade Soft Tissue Sarcomas - a Prospective, Comparative Study
Brief Title: Low-dose Computer Tomography in Follow-up of Soft Tissue Sarcomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Finnish Cancer Society (Unknown)
Responsible Party: Principal Investigator, Mika Sampo, Senior Consultant, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RADPOS1
Record Dates: First submitted 2023-03-30; First posted 2023-04-14 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Sarcoma,Soft Tissue
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chest x-ray and ultra-low-dose computed tomography (Experimental)
  Interventions: Diagnostic Test: ultra-low-dose computed tomography

INTERVENTIONS:
Diagnostic Test: ultra-low-dose computed tomography — 7 ultra-low-dose computed tomography imaging

SUMMARY:
The goal of this interventional study is to compare sensitivity of regular chest x-ray to ultra-low-dose computed tomography to find pulmonary relapse in follow-up of soft tissue sarcoma. The main question[s] it aims to answer are:

* Is ultra-low-dose computed tomography more sensitive than regular chest x-ray to find pulmonary relapse?
* Does ultra-low-dose computed tomography detect the most fast-growing pulmonary metastases earlier than regular chest x-ray?

Participants will have seven ultra-low-dose computed tomography imagings in addition to simultaneous routine protocol of chest x-rays. Participants therefore work as their own controls.

DETAILED DESCRIPTION:
After primary treatment with curative intent for soft tissue sarcoma, patients fulfilling the inclusion criteria and giving informed consent are enrolled. In study protocol patients have their regular chest x-ray once in two months plus ultra-low-dose computed tomography imaging is repeated seven times during the first two years of follow-up. After two years patients without detectable metastases continue in regular follow-up program. The aims of this prospective comparative study are to investigate whether ultra-low-dose computed tomography is more accurate than chest x-ray in soft tissue sarcoma and especially whether the most fast-growing pulmonary metastases could be detected earlier.

ELIGIBILITY:
Inclusion Criteria:

* primary high grade soft tissue sarcoma with no metastases at diagnoses or during treatment and treatment with curative intent.

Exclusion Criteria:

* metastases at diagnoses or during treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with pulmonary relapse detected by ultra-low-dose CT performed according to a pre-defined schedule | 2 years
Number of patients with pulmonary relapse detected by chest x-ray performed according to a pre-defined schedule | 2 years
Number of patients with pulmonary relapse by symptoms | 2 years
  Pulmonary relapse based on patient-reported symptoms leading to positive finding in x-ray and or conventional chest CT between two control imaging rounds.

CONTACTS AND LOCATIONS:
Overall Officials: Mika Sampo, MD PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital Comprehensive Cancer Center, Helsinki, Valitse Alue, Osavaltio Tai Maakunta, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Treasure T, Fiorentino F, Scarci M, Moller H, Utley M. Pulmonary metastasectomy for sarcoma: a systematic review of reported outcomes in the context of Thames Cancer Registry data. BMJ Open. 2012 Oct 8;2(5):e001736. doi: 10.1136/bmjopen-2012-001736. Print 2012. PMID 23048062
- [Background] Nevala R, Jaamaa S, Tukiainen E, Tarkkanen M, Rasanen J, Blomqvist C, Sampo M. Long-term results of surgical resection of lung metastases from soft tissue sarcoma: A single center experience. J Surg Oncol. 2019 Aug;120(2):168-175. doi: 10.1002/jso.25504. Epub 2019 May 27. PMID 31134646
- [Background] Dammerer D, VAN Beeck A, Schneeweiss V, Schwabegger A. Follow-up Strategies for Primary Extremity Soft-tissue Sarcoma in Adults: A Systematic Review of the Published Literature. In Vivo. 2020 Nov-Dec;34(6):3057-3068. doi: 10.21873/invivo.12140. PMID 33144410
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] Katsura M, Matsuda I, Akahane M, Yasaka K, Hanaoka S, Akai H, Sato J, Kunimatsu A, Ohtomo K. Model-based iterative reconstruction technique for ultralow-dose chest CT: comparison of pulmonary nodule detectability with the adaptive statistical iterative reconstruction technique. Invest Radiol. 2013 Apr;48(4):206-12. doi: 10.1097/RLI.0b013e31827efc3a. PMID 23344517
- [Background] Kaasalainen T, Makela T, Kelaranta A, Kortesniemi M. The Use of Model-based Iterative Reconstruction to Optimize Chest CT Examinations for Diagnosing Lung Metastases in Patients with Sarcoma: A Phantom Study. Acad Radiol. 2019 Jan;26(1):50-61. doi: 10.1016/j.acra.2018.03.028. Epub 2018 Apr 30. PMID 29724675
- [Background] Puri A, Gulia A, Hawaldar R, Ranganathan P, Badwe RA. Does intensity of surveillance affect survival after surgery for sarcomas? Results of a randomized noninferiority trial. Clin Orthop Relat Res. 2014 May;472(5):1568-75. doi: 10.1007/s11999-013-3385-9. Epub 2013 Nov 19. PMID 24249538
- [Derived] Salminen S, Jaamaa S, Nevala R, Sormaala MJ, Koivikko M, Tukiainen E, Repo J, Blomqvist C, Sampo M. Ultra-low-dose computed tomography and chest X-ray in follow-up of high-grade soft tissue sarcoma-a prospective comparative study. Sci Rep. 2024 Mar 26;14(1):7181. doi: 10.1038/s41598-024-57770-z. PMID 38531939